CLINICAL TRIAL: NCT05344170
Title: A Randomised, Double-blind, Placebo-controlled, Single-dose, Crossover, Pilot Study Investigating the Effects of Cannabinol (CBN) 30 mg and 300 mg on Sleep Architecture and Next-day Function in Insomnia Disorder
Brief Title: Cannabinol Use in Patients With Insomnia Disorder
Acronym: CUPID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112/2021-08-907
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-05

CONDITIONS: Insomnia Disorder
Keywords: cannabinol; CBN; cannabinoid; medicinal cannabis; primary insomnia; chronic insomnia disorder; sleep architecture; wake after sleep onset; polysomnography; next-day function; randomised controlled trial; placebo-controlled; crossover; double-blinded
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cannabinol

STUDY DESIGN:
Intervention Model Description: Single site allocation: Randomised Intervention model: Crossover Masking: Double-blind (participant, investigator) Primary purpose: Pilot
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind: Eligible participants will be assigned to one of six possible treatment orders using a pre-populated randomisation schedule. Study staff (including the study investigators, the clinical trials coordinator and the study medical officer) and the participants will be blinded. Allocation concealment will be managed by the trial epidemiologist and drug distributor who will not have any contact with participants or involvement in day-to-day trial activities. Traditional polysomnographic (PSG) measures will be scored by a PSG technician who will not be aware of participant treatment, nor will they meet the participant. The study drug and matched placebo are expected to be identical in their visual appearance, taste, or smell. A mint-flavoured lozenge will be administered immediately prior to the study drug to mask any possible differences in taste.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30 mg Cannabinol (CBN) (Experimental): Single fixed dose administered 2 hours prior to habitual sleep onset.
  Interventions: Drug: 30 mg Cannabinol (CBN)
- 300 mg Cannabinol (CBN) (Experimental): Single fixed dose administered 2 hours prior to habitual sleep onset.
  Interventions: Drug: 300 mg Cannabinol (CBN)
- Placebo (Placebo Comparator): Single fixed dose administered 2 hours prior to habitual sleep onset.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 30 mg Cannabinol (CBN) — Participants will receive a 2 mL oral dose of 'ECS 310' (1.5%), an oral formulation of CBN (15 mg/mL) suspended in medium chain triglycerides (MCT) oil.
  Other Names: ECS 310 (1.5%)
  Arms: 30 mg Cannabinol (CBN)
Drug: 300 mg Cannabinol (CBN) — Participants will receive a 2 mL oral dose of 'ECS 310' (15%), an oral formulation of CBN (150 mg/mL) suspended in medium chain triglycerides (MCT) oil.
  Other Names: ECS 310 (15%)
  Arms: 300 mg Cannabinol (CBN)
Drug: Placebo — Participants will receive a 2 mL oral dose of placebo. Placebo contains the same excipient, medium chain triglycerides (MCT) oil, as the investigational products but does not contain cannabinoids.
  Arms: Placebo

SUMMARY:
This study aims to investigate the acute effects of cannabinol (CBN) 30 mg and 300 mg, versus placebo, on sleep architecture and next-day functioning in adults aged 25-65 years with chronic insomnia disorder.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, three-arm, crossover, single-centre, proof-of-concept study in twenty participants with chronic insomnia disorder (as per clinician diagnosis and Insomnia Severity Index [ISI] Score ≥15). Across three overnight treatment sessions, participants will receive single dose oral liquid 30 mg cannabinol (CBN), 300 mg CBN, and matched placebo. Participants will undergo overnight sleep assessment using in-laboratory polysomnography (PSG) to examine CBN-related changes to sleep parameters; and various objective and subjective measures of sleep and next-day neurobehavioral function. Each treatment session will be separated by the two-week washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Between 25 - 65 years of age
2. Insomnia Severity Index (ISI) score ≥ 15 at eligibility screening
3. Insomnia disorder (symptoms occurring at least 3 times per week and present for longer than 3 months) as determined by the study physician
4. Ability to take oral medication
5. Provision of signed and dated informed consent form
6. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

1. Medical condition or medication that is the cause of the insomnia disorder as determined by the study physician
2. Known hypersensitivity to cannabis or cannabinoid products (including if this becomes evident during the trial)
3. Reported use of cannabis or cannabinoid products within the past 3 months as confirmed by at least one negative urine drug screen (UDS) (or at the study physician's discretion)
4. Sleep apnoea (defined as Apnoea Hypopnea Index [AHI] > 15 and Oxygen Desaturation Index [ODI]>10) as confirmed by polysomnography at screening
5. Sleep-related movement disorder as determined by the study physician
6. Delayed or advanced sleep phase syndrome (based on actigraphy and sleep diary) as confirmed during screening
7. Any medical condition that produces an abnormal EEG (i.e., epilepsy, brain injury)
8. Clinically relevant cardiovascular abnormalities as determined by the study physician and a 12-lead electrocardiogram (ECG) at screening
9. Shift work or trans meridian travel (two time zones) within the last month
10. History of major psychiatric disorder in the past 12 months at the study physician's discretion, except clinically managed mild depression and/or anxiety
11. History of suicide attempt or current suicide ideation (score greater than 1 on Q9 of the Patient Health Questionnaire [PHQ-9])
12. Pregnancy or lactating. Female participants are required to complete a urine pregnancy test at screening and treatment sessions and all participants are instructed to use a reliable form of contraception throughout the study duration
13. History of drug or alcohol dependency or abuse within approximately the past 2 years
14. Use of CNS-active drugs (cannabis, amphetamines, cocaine, antidepressants, opioids, benzodiazepines) in the past 3 months as confirmed by a positive urine drug test at screening or at the study physician's discretion
15. Use of medications that may have a clinically significant impact upon the metabolism and excretion of cannabinoids as determined by the study physician (e.g., CYP450 enzyme inducers/inhibitors
16. Excessive caffeine use that in the opinion of the study physician contributes to the participant's insomnia disorder, or the inability to abstain from caffeine use 24 hours prior to each overnight sleep study
17. Inability to refrain from alcohol consumption 24 hours prior to each overnight sleep study
18. Individuals with nicotine dependence (i.e., daily smokers)
19. Medical conditions that result in frequent need to get out of bed (e.g., sleep walking, nocturia)
20. Psychological or behavioural treatment for insomnia disorder, including cognitive behavioural therapy for insomnia, within 3 months before screening (excluding sleep hygiene advice)
21. Occupational or judicially ordered drug screening
22. Has held an unrestricted driving license < 1 year
23. Cannot speak English fluently

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Wake After Sleep Onset (WASO) | Night 1
  WASO measured in minutes using in-laboratory overnight polysomnography, from the first epoch after lights out until the last epoch, scored as any stage of sleep by an experienced polysomnographic technician in accordance with American Academy of Sleep Medicine (AASM) 2020 Sleep Scoring criteria (Version 2.6). Comparisons between each CBN dose versus placebo.

SECONDARY OUTCOMES:
Traditional sleep staging | Night 1
  Proportion of the sleep opportunity scored at the 5 stages (wake, and N1, N2, N3, and REM sleep) between lights out and lights on, measured using overnight in-laboratory polysomnography, scored by a polysomnography technician in accordance with AASM Sleep Scoring criteria. Comparisons between each CBN dose versus placebo.
Sleep Onset Latency (SOL) | Night 1
  SOL measured in minutes using in-laboratory polysomnography, calculated from the time of lights out to the first sleep epoch as scored by a polysomnographic technician in accordance with AASM Sleep Scoring criteria. Comparisons between each CBN dose versus placebo.
Absolute Electroencephalographic (EEG) Power During Non-Rapid Eye Movement (NREM) Sleep. | Night 1
  Spectral power of delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges between treatment arms. Power spectral analysis will be applied to EEG signals from polysomnography after artefacts are detected and removed. Comparisons between each CBN dose versus placebo.

OTHER OUTCOMES:
Sleep Spindles During Non-Rapid Eye Movement (NREM) Sleep (Tertiary outcome) | Night 1
  Sleep spindle and slow oscillation events in NREM sleep from in-laboratory overnight polysomnography. A sleep spindle and slow oscillation detection algorithm will be applied to electroencephalography (EEG) signals from polysomnography after artefacts are detected and removed. Comparisons between each CBN dose versus placebo.
Electroencephalogram (EEG) Arousal Index (Tertiary outcome) | Night 1
  Number of cortical arousals captured via the electroencephalogram per hour of sleep scored by the polysomnographic technician on the polysomnogram in accordance with AASM Sleep Scoring criteria. Comparisons between each CBN dose versus placebo.
Absolute Electroencephalography (EEG) Power During Rapid Eye Movement (REM) Sleep (Tertiary outcome) | Night 1
  Spectral power of delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges between treatment arms. Power spectral analysis will be applied to EEG signals from polysomnography after artefacts are detected and removed. Comparisons between each CBN dose versus placebo.
Next day post-wake subjective sleep evaluation (LSEQ) (Tertiary outcome) | Morning after drug administration
  LSEQ score. LSEQ scores range from 0-100, with higher scores indicating better subjective experience. Assessed within 1 h after wake (comparison between each CBN dose versus placebo).
Next day post-wake subjective sleep evaluation (RCSQ) (Tertiary outcome) | Morning after drug administration
  RCSQ score. RCSQ scores range from 0-100, with higher scores indicating better subjective experience. Assessed within 1 h after wake (comparison between each CBN dose versus placebo).
Standard Deviation of Lateral Position (SDLP) During Next-day Post-Wake Simulated Drive (Safety outcome) | Morning after drug administration
  SDLP ("weaving") is measured across the 'standard', 'car following', and 'divided attention' sub-sections of a ~30 minute simulated driving task. Assessed within 2 h after wake (comparison between each CBN dose versus placebo).
Speed During Next-day Post-Wake Simulated Drive (Safety outcome) | Morning after drug administration
  Average speed and standard deviation of speed is measured across the 'standard' and 'divided attention' sub-sections of a ~30 minute simulated driving task. Assessed within 2 h after wake (comparison between each CBN dose versus placebo).
Distance Headway During Next-day Post-Wake Simulated Drive (Safety outcome) | Morning after drug administration
  Average distance headway (i.e., distance between the driver's vehicle and vehicle immediately in front) and standard deviation of distance headway is measured across the 'car following' sub-section of a ~30-minute simulated driving task. Assessed within 2 h after wake at both treatment sessions (comparison between each CBN dose versus placebo).
Subjective Mood Evaluation (Safety outcome) | Immediately after and morning after drug administration
  The Abbreviated Profile of Mood States (POMS) consists of 40 items measuring domains of 'tension', 'depressed', 'anger', 'vigour', 'fatigue', and 'concentration'. Participants respond to each item using 5-point Likert scales ranging from 0 (Not at all) to 4 (Extremely). A total mood disturbance score is calculated by summing negative domains and subtracting positive domains. Administered pre and post drug administration, as well as next-day (comparison between each CBN dose versus placebo).
Subjective Drug Effects (Safety outcome) | Immediately after and morning after drug administration
  The Drug Effects Questionnaire (DEQ) assesses the extent to which participants feel a drug effects, feel high, like the effects, dislike the effects, want more of the substance, and feel sedated, on self-rating 100mm visual analogue scales. A total mood disturbance score is calculated by summing negative domains and subtracting positive domains. Administered pre and post drug administration, as well as next-day (comparison between each CBN dose versus placebo).
Postural sway (Safety outcome) | Immediately after and morning after drug administration
  Centre-of-pressure (COP) during computerised static posturography. Administered pre and post drug administration, as well as next-day (comparison between each CBN dose versus placebo).
Behavioural Alertness and Reaction Time (Safety outcome) | Morning after drug administration
  Psychomotor Vigilance Test (PVT) is administered twice the next-day (comparison between each CBN dose versus placebo).
Overnight Declarative Memory Consolidation (Safety outcome) | Morning after drug administration
  Word pair recall scores measured using the computerised Word Pairs Task (WPT). Administered pre-drug administration and next-day (comparison between each CBN dose versus placebo).
Overnight Procedural Memory Consolidation (Safety outcome) | Morning after drug administration
  Motor sequence learning measured using the computerised Finger Tapping Task (FTT). Administered pre-drug administration and next-day (comparison between each CBN dose versus placebo).
Resting Wake Electroencephalography (EEG) Power After Sleep (Post-Wake Effects) (Safety Outcome) | Morning after drug administration
  Resting wake EEG power during the Karolinska Drowsiness Test (KDT) upon wake: delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges. Power spectral analysis is applied to EEG signals from polysomnography, after artefacts are detected and removed. Comparison between each CBN dose versus placebo.
Subjective sleepiness after sleep | Morning after drug administration
  The Karolinska Sleepiness Scale (KSS) is a 10-item measure of subjective drowsiness. Participants respond to each item using a 9-point Likert scale ranging from 1 (Extremely alert) to 9 (Extremely sleepy). Higher scores are indicative of increased drowsiness. The KSS will be collected in accordance with the KDT protocol but will not be analysed due to insufficient statistical power.
Resting Wake Electroencephalography (EEG) Power Before Sleep (Acute Effects)(Exploratory outcome) | Immediately after drug administration
  Resting wake EEG power during the KDT prior to sleep: delta (1-4.5 Hz), theta (4.5-8 Hz), alpha (8-12 Hz), sigma (12-15 Hz), beta (15-25 Hz), and gamma (25-40 Hz) frequency ranges. Power spectral analysis is applied to EEG signals from polysomnography, after artefacts are detected and removed. Comparison between each CBN dose versus placebo.
Subjective sleepiness after sleep (acute effects) (Exploratory outcome) | Immediately after drug administration
  The KSS is a 10-item measure of subjective drowsiness. Participants respond to each item using 9-point Likert scales ranging from 1 (Extremely alert) to 9 (Extremely sleepy). Higher scores are indicative of higher drowsiness. The KSS will be collected in accordance with the KDT protocol but will not be analysed due to insufficient statistical power.
Plasma cannabinoid concentrations (Exploratory outcome) | Immediately after and morning after drug administration
  Presence of cannabinoids (CBN, delta-9-tetrahydrocannabinol [THC], and cannabidiol [CBD]) (e.g., 11-OH-CBN, 11-COOH-CBN, 11-OH-THC, 11-COOH-THC, 7-OH-CBD, 7-COOH-CBD), and endocannabinoids and related molecules (e.g., 2-Arachidonoylglyceroland anandamide) and their metabolites in plasma samples.
Urinary cannabinoid concentrations (Exploratory outcome) | Immediately after and morning after drug administration
  Presence of cannabinoids (CBN, THC, and CBD) and their metabolites (11-OH-CBN, 11-COOH-CBN, 11-OH-THC, 11-COOH-THC, 7-OH-CBD, 7-COOH-CBD) in urine samples.
Salivary cannabinoid concentrations (Exploratory outcome) | Immediately after and morning after drug administration
  Presence of cannabinoids (THC, CBN) and their metabolites (11-OH-CBN, 11-COOH-CBN, 11-OH-THC, 11-COOH-THC) in saliva samples.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Hoyos, MPH, PhD, Principal Investigator — Woolcock Institute of Medical Research; Brendon Yee, MBChB, FRACP, FCCP, PhD, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Glebe, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable IPD will be shared upon reasonable request to the Chief Investigators.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Non-identifiable IPD will become available one year after the Actual Study Completion Date and will be available for 10 years.
Access Criteria: Individual participant level meta-analyses of congruent studies

REFERENCES:
- [Derived] Lavender I, McCartney D, Marshall N, Suraev A, Irwin C, D'Rozario AL, Gordon CJ, Saini B, Grunstein RR, Yee B, McGregor I, Hoyos CM. Cannabinol (CBN; 30 and 300 mg) effects on sleep and next-day function in insomnia disorder ('CUPID' study): protocol for a randomised, double-blind, placebo-controlled, cross-over, three-arm, proof-of-concept trial. BMJ Open. 2023 Aug 23;13(8):e071148. doi: 10.1136/bmjopen-2022-071148. PMID 37612115